CLINICAL TRIAL: NCT04034654
Title: Behavioral Assessment of Preschool Children Who Had Undergone General Surgery in Early Infancy
Brief Title: Behavioral Assessment of Operated Preschool Children
Acronym: BASIS
Status: Completed | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Danguole C Rugyte, Professor, MD PhD, Lithuanian University of Health Sciences
Other Study IDs: P1-BE-2
Record Dates: First submitted 2019-01-30; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Child Behavior; Anesthesia; Peri-operative Injury
Keywords: preschool child; behavior; anesthesia; surgery
MeSH Terms: conditions — Child Behavior; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionaire — Child behavior checklist is a questionaire, designed to evaluate 1.5-5 years old child's behavior. The checklist is filled out by parents/caregivers.
  Other Names: Child behavior checklist

SUMMARY:
This study will investigate the behavior of preschool children who had undergone general surgery during early infancy and will correlate the behavioral outcomes with clinical perioperative variables.

DETAILED DESCRIPTION:
Several epidemiologic and observational studies found the relation between surgery in childhood and neurodevelopmental features in later life. However, these studies are criticized for retrospective design, non homogenous population, social confounders, diversity of surgical procedures and anesthetic management.

Monitoring of neurological function has become standard during surgical procedures at risk for neuronal injury (e.g. cardiac surgery). There is also some data on possible predictive value of certain methods of neuromonitoring (such as cerebral near infrared spectroscopy (NIRS)) for neurodevelopmental outcome.

General neonatal/infant surgery and the whole perioperative period carry the risk of significant physiologic disturbances, which may affect cerebral perfusion, oxygenation or metabolism. This study is the continuum of prospective observational trial, which investigated the value of the neuromonitoring measures in neonates and young infants undergoing general surgery. The present study will apply the behavioral assessment of these patients who are now between 2 and 5 years of age.

ELIGIBILITY:
Inclusion Criteria:

* children, who had undergone general surgery for congenital anomalies or disease from birth until 93 days of age at a single University hospital
* general anesthesia with inhalational anesthetic was applied during surgery
* artificial lung ventilation was applied during anesthesia
* NIRS values were recorded throughout anesthesia
* serum concentrations of brain specific proteins were obtained during perioperative period

Exclusion Criteria:

* children, who had undergone cardiac, neurosurgical, ear, nose and throat or eye surgery from birth until 93 days of age
* general anesthesia without tracheal intubation was applied
* local or combined local/general anesthesia was applied

Ages: 18 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children, aged 1.5-5 years, who had undergone general abdominal, thoracic, genitourinary surgery until 93 days of life in a single University hospital and were given standard inhalational general anesthesia with tracheal intubation and measures for neuromonitoring such as cerebral NIRS and measurement of brain specific proteins during perioperative period was applied.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
abnormal behavioral outcome as assessed by CBCL | 2 to 5 year after surgery
  the number of children with one or more abnormal behavioral domains

CONTACTS AND LOCATIONS:
Overall Officials: Danguole Rugyte, MD PhD, Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania